CLINICAL TRIAL: NCT03094871
Title: FACE-PC: Family-Centered Care for Older Adults With Depression and Chronic Medical Conditions in Primary Care
Acronym: FACE-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-23224
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Chronic Medical Conditions; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): FACE-PC comprises 3 weekly and 2 bi-weekly sessions (total 5 sessions), delivered by a bachelors' prepared nurse care manager (CM) over 8 weeks. Over the five sessions, the nurse care manager will (1) review the patient medical history and set health goals for depression and chronic condition with the dyad, (2) review all medication, the level of adherence, challenges and facilitating factors of adherence, (3) deliver brief behavioral activation therapy.
  Interventions: Behavioral: FACE-PC
- Enhanced usual care group (No Intervention): Participants in this group will receive a typical primary care enhanced with reporting of their depression status and their goal for medical condition to their PCP for 8 weeks. Upon enrolment, a research nurse will review the patient medical history and identify goals for depression and a chronic condition with the dyad.

INTERVENTIONS:
Behavioral: FACE-PC
  Arms: Intervention group

SUMMARY:
Comorbid depression and multiple medical conditions in older adults are a serious public health problem. As an important facilitator of health-related activities, families are already involved in various aspects of self-management of chronic disease in older adults. Despite the benefits they provide, informal caregiving activities currently are organized outside the medical system, which potentially creates redundant or misaligned efforts.The purpose of the mentored research is to examine the feasibility and acceptability of the FACE-PC, a theory-driven, multi- component, technology-assisted interdisciplinary team-based care model that systematically involves family in chronic disease management. It aims to optimize the patient and family's collective ability to self-manage chronic disease.

DETAILED DESCRIPTION:
Comorbid depression and multiple medical conditions in older adults are a serious public health problem. As an important facilitator of health-related activities, families are already involved in various aspects of self-management of chronic disease in older adults. Despite the benefits they provide, informal caregiving activities currently are organized outside the medical system, which potentially creates redundant or misaligned efforts.The purpose of the mentored research is to examine the feasibility and acceptability of the FACE-PC, a theory-driven, multi- component, technology-assisted interdisciplinary team-based care model that systematically involves family in chronic disease management. It aims to optimize the patient and family's collective ability to self-manage chronic disease.

ELIGIBILITY:
Inclusion Criteria for Patient:

* 60 years of age or older
* Receives primary care
* PHQ-9 score ≥ 5
* Must have at least one medical condition actively managed at the study site.

Inclusion Criteria for Family:

* Age 18 or older
* Identified as family by the patient
* Has a minimum of twice weekly total of 4 hour face-to face contact with the patient
* Is willing and available to participate in the study;
* Has access to internet.

Exclusion Criteria for Patient:

* Inability to understand screening and assessment questions
* Montreal Cognitive Assessment Scores <18
* Known diagnosis of a severe chronic mental illness such as schizophrenia
* Meeting the criteria for bipolar disorder or schizophrenia in PRIME-MD
* Deemed to be a danger to self or others that may require treatment outside a primary care setting.

Exclusion Criteria for Family:

* Institutionalized at the time of study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in Mood assessed with Patient Health Questionnaire | at baseline, 2-months post-intervention, and 5-months follow-up
  Patient Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mijung Park, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No